CLINICAL TRIAL: NCT00998504
Title: Effect of resVida on Fat Oxidation and Mitochondrial Biogenesis in Healthy Obese Subjects
Brief Title: resVida and Fat Oxidation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry); Top Institute Food and Nutrition (Other)
Responsible Party: Silvie Timmers, MSc, Top Institute Food and Nutrition
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MEC 09-3-039
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2011-03-18 (Estimated); Status verified 2011-03

CONDITIONS: Obesity
Keywords: impaired fat oxidation; fat accumulation; mitochondrial dysfunction; mitochondrial biogenesis
MeSH Terms: conditions — Obesity; Mitochondrial Diseases | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): starch pill
  Interventions: Dietary Supplement: placebo
- resVida (Active Comparator): synthetic pill containing 75 mg of resveratrol
  Interventions: Dietary Supplement: resVida

INTERVENTIONS:
Dietary Supplement: resVida — resVida or placebo will be given for 30 days, twice daily. One pill, which contains 75 mg of resVida, will be provided with lunch, and the other pill will be provided with diner. So in total, 150 mg/day will be given.
  Other Names: resveratrol
  Arms: resVida
Dietary Supplement: placebo — resVida or placebo will be given for 30 days, twice daily. One pill, which contains 75 mg of resVida, will be provided with lunch, and the other pill will be provided with diner. So in total, 150 mg/day will be given.
  Arms: placebo

SUMMARY:
There is now a general consensus that the combination of excessive energy intake and a low capacity to oxidize fat will lead to muscular fat accumulation and insulin resistance. It is known for many years that physical exercise is the most powerful treatment to combat insulin resistance, but it is also known that it is difficult to get people to exercise. A major breakthrough has come from the nutrition field, with the finding that resveratrol, a natural polyphenolic compound, could serve as an "exercise mimetic" by protecting mice from many detrimental effects of diet-induced obesity. Therefore the researchers would like to investigate if resVida can increase skeletal muscle mitochondrial function and fat oxidative capacity in obese subjects. The researchers hypothesize that an increased mitochondrial function together with an increased intrinsic activity will lead to a better control of fatty acid handling in muscle, upon a high-fat challenge.

ELIGIBILITY:
Inclusion Criteria:

* male sex
* age 45-65 years
* body fat percentage > 25%, BMI 30-35 kg/m2
* sedentary
* stable dietary habits
* willingness to abstain from ingestion of resveratrol-containing foods
* healthy

Exclusion Criteria:

* female sex
* unstable body weight (weight gain or loss > 3 kg in the last three months)
* total body fat percentage < 25%
* fasting plasma glucose > 6.1 mmol/l
* hemoglobin < 7.8 mmol/l
* engagement in programmed exercise > 2 hours total per week
* impaired kidney and/ or liver function
* first- or second-degree family member with type 2 diabetes mellitus
* any medical condition requiring treatment and/ or medication use
* intake of dietary supplements except vitamins and minerals
* unwilling to restrict high-resveratrol containing foods
* current alcohol consumption > 20 grams/day
* participation in another biomedical study within 1 month before the screening visit
* a contraindication to MRI scanning. These contraindications include patients with the following devices:
* central nervous system aneurysm clips
* implanted neural stimulator
* implanted cardiac pacemaker or defibrillator
* cochlear implant
* insulin pump
* or metal containing corpora aliena in the eye or brains

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
difference in fat oxidation between resVida and placebo treated group | 9 months

SECONDARY OUTCOMES:
difference in mitochondrial biogenesis, function, and lipolysis in adipose and skeletal muscle tissue between resVida and placebo treated group | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Silvie Timmers, MSc, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Knop FK, Konings E, Timmers S, Schrauwen P, Holst JJ, Blaak EE. Thirty days of resveratrol supplementation does not affect postprandial incretin hormone responses, but suppresses postprandial glucagon in obese subjects. Diabet Med. 2013 Oct;30(10):1214-8. doi: 10.1111/dme.12231. Epub 2013 Jun 7. PMID 23663119